CLINICAL TRIAL: NCT05721794
Title: Comparative Accuracy of Transperineal Ultrasound (TPUS) Versus Magnetic Resonance Imaging (MRI) for the Assessment of Perianal Fistulae in Patients With Crohn's Disease (CD): a Prospective Observational Longitudinal Cohort Study
Acronym: TPUS-MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Mariangela Allocca, gastroenterologist physician, IRCCS San Raffaele
Other Study IDs: TPUS-MRI
Record Dates: First submitted 2023-01-27; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Crohn Disease; Perianal Fistula
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: A multicentric prospective observational longitudinal cohort study. — Observational study on the accuracy of TPUS and MRI in the investigation of perianal fistulae in CD patients.

SUMMARY:
Crohn's disease (CD) is a life-long chronic inflammatory bowel disease (IBD) that may affect any site of the gastrointestinal tract, most frequently the ileum and colon. It is characterized by transmural inflammation and it can lead to strictures, due to activation of reparation of inflamed tissues and consequent fibrosis, or penetrating lesions, such as fistulas, between two different intestinal tracts or between intestine and surrounding organs. Fistula occurrence can lead to formation of abdominal or pelvic abscesses. Such complications cause intestinal damage and usually require surgery, leading to disability, impairment of patients' quality of life, with significant impact on direct and indirect health-care costs

DETAILED DESCRIPTION:
The investigators aim to conduct a multicentric pilot prospective observational study on the accuracy of TPUS and MRI in the investigation of perianal fistulae in CD patients. Fifty adult patients with confirmed diagnosis of Crohn's disease and perianal fistulae will be enrolled by five international centres between June 2022 and June 2023.

According to the observational nature of the study, all the visits and procedures described below will be performed according to the diagnostic and therapeutic assignment required by clinical practice for the patients under study. TPUS and MRI are normally performed by clinical practice. The choice of treatment for the cure of the fistula (e.g. medical and / or surgical treatment) will be made by the referring physicians according to the international ECCO guidelines. Therefore, the choice of assigning the patient to the diagnostic and therapeutic procedures deemed most appropriate for each case is completely independent of the study.

Subjects will undergo both TPUS and pelvic MRI at baseline as for clinical practice. After radiological and ultrasound evaluation, subjects will be treated according to international ECCO guidelines. In particular, patients will undergo seton insertion and 2 weeks later they will start biologics at the discretion of the gastroenterologist in according with international guidelines . Surgical closure with the advancement flap (AF) or Ligation of the Intersphincteric Fistula Tract (LIFT) procedure will occur 8-12 weeks after seton placement, with seton removal during surgical closure. The choice of surgical technique will be at the discretion of the surgeon. Finally patients will undergo both TPUS and pelvic MRI after 12 months as for clinical practice.

TPUS findings will be compared with those of the standard MRI to assess perianal disease activity. For that purpose, the investigators will:

1. Identify 50 CD patients with perianal fistulae. Those patients will undergo both standard pelvic MRI and TPUS.
2. Treat all patients with perianal fistulae according to international guidelines (e.g., medical and/or surgical treatment).
3. Monitor all patients included according to the scheduled follow-up to evaluate the value of TPUS findings in assessing perianal disease evolution.

Fistulae identified will be classified according to the MAGNIFI-CD Activity Index, a validated score ranging from 0 to 25. For both TPUS and MRI the positive value, indicating the presence of the fistula, is considered for a MAGNIFI-CD>6. It evaluates several items including the number of fistulas, length of fistulas, extension, presence of inflammatory mass, dominant features, and hyperintensity on post-contrast T1-weighted images. The investigators will calculate the MAGNIFI-CD also with the TPUS and they will evaluate if the results of the score obtained with the ultrasound are correlated to those obtained with the MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >18 years
2. Confirmed diagnosis of Crohn's disease.
3. Clinical suspicion of perianal fistulae (e.g., perianal pain or swelling, drainage of pus, stool or stool from cutaneous fistula opening, and signs and symptoms of sepsis)
4. Able to understand and sign an informed consent form

Exclusion Criteria:

1. Controindications to MRI
2. Severe comorbidities that limit the performance of MRI and TPUS
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 adult patients with confirmed diagnosis of Crohn's disease and suspicion of perianal fistulae will be enrolled in the study. Number and length of fistulae will be evaluated through MRI and TPUS. In addition, the response to treatment, defined as rate of fistula closure will also be evaluated with both techniques
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-06-06 (Estimated); Study Completion 2024-06-06 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of perianal fistulae through the MAGNIFI-CD index (by TPUS) and the standard MAGNIFI-CD index (by MRI) | 1 year
  To compare the accuracy of the TPUS versus pelvic MRI in assessing perianal fistulae in CD patients. Accuracy is defined as the ability to identify perianal fistulae

SECONDARY OUTCOMES:
Rate of fistula closure, determined by the clinician, at 12 months. | 1 year
  To compare the accuracy of the TPUS versus pelvic MRI in evaluating response to treatment in CD patients with fistulae

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Allocca, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Mariangela Allocca, Milan, Italy